CLINICAL TRIAL: NCT03795753
Title: Determining the Benefits of Improving Communication in BPAP/CPAP Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nancy Abbey Collop, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00097529
Record Dates: First submitted 2018-12-28; First posted 2019-01-08 (Actual); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-08

CONDITIONS: Positive-Pressure Respiration; Communication
Keywords: Emphysema; Chronic obstructive pulmonary disease; Obstructive sleep apnea
MeSH Terms: conditions — Communication; Emphysema; Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- F2S Communicator (Experimental): The F2S Communication System is a communication aid for use with a noninvasive ventilation (NIV) mask covering at least the mouth. It is a two-component system consisting of (1) a disposable, single patient use patch and signal cable and (2) a reusable communicator with power cable.The non-invasive aid for patients receiving BPAP/CPAP therapy delivers communication between the patient and medical personnel.
  Interventions: Device: F2S Communicator
- Non-functioning Communicator (Sham Comparator): Non-functioning study communication device is used.
  Interventions: Other: Non-functioning Communicator

INTERVENTIONS:
Device: F2S Communicator — The communicator will be attached to the BPAP/CPAP mask. The study coordinator will ENABLE the communicator. A list of single words and 5-word through 15-word sentences will be provided to the patient. Each single word may be read aloud up to two times. The partner must then select the read word out of a list of twelve possible words. Each sentence may be read aloud up to two times. The partner must transcribe each sentence on a standardized form. A survey will be provided to evaluate the "mask on, communicator on" period.
  Other Names: BPAP/CPAP communicator
  Arms: F2S Communicator
Other: Non-functioning Communicator — The communicator will be attached to the BPAP/CPAP mask. The study coordinator will DISABLE the communicator. A list of single words and 5-word through 15-word sentences will be provided to the patient. Each single word may be read aloud up to two times. The partner must then select the read word out of a list of twelve possible words. Each sentence may be read aloud up to two times. The partner must transcribe each sentence on a standardized form. A survey will be provided to evaluate the "mask on, communicator on" period.
  Arms: Non-functioning Communicator

SUMMARY:
The purpose of this study is to determine the effectiveness of a non-invasive communication aid for BPAP/CPAP masks. This study also looks to determine the potential impact of the device on patients with obstructive sleep apnea (OSA) and the individuals that interact with the device.

DETAILED DESCRIPTION:
Noninvasive positive pressure ventilation (NIPPV) is a crucial tool used to treat respiratory distress and failure, especially when patients have acute worsening (also called exacerbations) of emphysema or chronic obstructive pulmonary disease (COPD). This study will randomize patients who use Noninvasive positive pressure ventilation (NIPPV) to a control (non-functioning) and intervention (functioning) device to determine how well speech can be understood while wearing the device.

The purpose of this study is to determine the effectiveness of a non-invasive communication aid for BPAP/CPAP masks. This study also looks to determine the potential impact of the device on patients with obstructive sleep apnea (OSA) and the individuals that interact with the device.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be receiving BPAP/CPAP therapy in the outpatient setting (e.g. clinics, sleep centers).

Exclusion Criteria:

* Intubated or have a tracheostomy.
* Vulnerable populations (children, pregnant women, decisionally impaired adults, and prisoners).
* Speech disabilities, reading disabilities, dyslexia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Collop, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong AI, Cheung PC, Zhang J, Cotsonis G, Kutner M, Gay PC, Collop NA. Randomized Controlled Trial of a Novel Communication Device Assessed During Noninvasive Ventilation Therapy. Chest. 2021 Apr;159(4):1531-1539. doi: 10.1016/j.chest.2020.09.250. Epub 2020 Oct 1. PMID 33011202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | F2S Communicator | Non-functioning Communicator
Started | 23 | 13
Completed | 23 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | F2S Communicator | Non-functioning Communicator | Total
Number analyzed (Participants) | 23 | 13 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (13.3) | 59.9 (17.1) | 57.03 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 4 | 17
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 13 | 36

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Single Word Selection (Proportion of Right Words From Total)
Description: Data will be collected using audio recording - accuracy of single word selection (spoken by patient -> selected by partner). The communicator will be attached to the BPAP/CPAP mask. A list of single words will be provided to the patient. Each single word may be read aloud by patient up to two times. The partner must then select the read word out of a list of twelve possible words.
Time Frame: Mask on-communicator on-20 minutes
Measure: Mean (Standard Deviation); unit: proportion of right words
Arm/Group | F2S Communicator | Non-functioning Communicator
Number analyzed (Participants) | 23 | 13
proportion of right words | 0.61 (0.13) | 0.35 (0.17)

2. Primary Outcome: Accuracy of Sentence Selection (Proportion of Right Sentences From Total)
Description: Data will be collected using audio recording - accuracy of sentence selection (spoken by patient -> transcribed by partner). The communicator will be attached to the BPAP/CPAP mask. A list of 5-word through 15-word sentences will be provided to the patient. Each sentence may be read aloud by patient up to two times. The partner must transcribe each sentence on a standardized form.
Time Frame: Mask on-communicator on-20 minutes
Measure: Mean (Standard Deviation); unit: proportion of sentence intelligibility
Arm/Group | F2S Communicator | Non-functioning Communicator
Number analyzed (Participants) | 23 | 13
proportion of sentence intelligibility | 0.76 (0.22) | 0.33 (0.25)

3. Secondary Outcome: Speech Transmission Index (STI)
Description: STI is a numeric representation measure of communication channel characteristics whose value varies from 0 = bad to 1 = excellent.On this scale, an STI of at least 0.5 is desirable for most applications.
Time Frame: Mask on with communicator on (20 min)
Population: A validated conversion for word/sentence accuracy and STI was not predetermined and the intent was to record at both the mask and the speaker. However, the conversion was not able to be determined and recording at the mask level was limited by the device. Thus, there is no effective comparator to calculate STI and this information is unavailable.
Arm/Group | F2S Communicator | Non-functioning Communicator
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Subjects That Found That the Device Significantly Improved Noninvasive Ventilation (NIV) Comfort
Description: Number of subjects that found that the device significantly improved noninvasive ventilation (NIV) comfort was calculated and reported. Assessment of noninvasive ventilation (NIV) comfort was conducted using Likert Scale Score on clarity of communication on a symmetric seven-level agree-disagree scale.
Time Frame: Mask on-communicator on-20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | F2S Communicator | Non-functioning Communicator
Number analyzed (Participants) | 23 | 13
Participants | 11 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | F2S Communicator | Non-functioning Communicator
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/13
Other Adverse Events (participants affected / at risk) | 0/23 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03795753/Prot_SAP_000.pdf